CLINICAL TRIAL: NCT04659200
Title: Thyroid Function Tests and the Status of Thyroid Autoantibodies in Hospitalized Covid-19 Patients and Their Relationship With White Blood Cells, Neutrophil / Lymphocyte Ratio, c Reactive Protein, Fibrinogen, Procalcitonin, Ferritin and D-dimer
Brief Title: Thyroid Function Tests and Status of Thyroid Autoantibodies in Covid-19 Patients
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Sabahattin Destek, Associate Professor, Bezmialem Vakif University
Other Study IDs: 06122020
Record Dates: First submitted 2020-12-07; First posted 2020-12-09 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: COVID-19 Infection; Thyroid Function Tests; Inflammation; Thyroid; Inflammatory Markers
MeSH Terms: conditions — COVID-19; Inflammation; Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid Disease Patient Group: Researchers evaluated serum thyrotropin, free triiodothyronine, free thyroxine hormones, thyroid peroxidase antibodies and anti-thyroglobulin antibodies in patients hospitalized for COVID-19 infection. The researchers evaluated the results of white blood cells, neutrophil / lymphocyte ratio, c reactive protein, fibrinogen, procalcitonin, ferritin, D-dimer in Covid-9 patients.
  Interventions: Diagnostic Test: Venous blood was collected for biochemistry testing.
- Covid-Free Control Group: Researchers evaluated the results of serum thyrotropin, free triiodothyronine, free thyroxine hormones, thyroid peroxidase antibodies and anti-thyroglobulin antibodies, white blood cells, neutrophil / lymphocyte ratio, c reactive protein, fibrinogen, procalcitonin, ferritin, D-dimer in the non-patient control group.
  Interventions: Diagnostic Test: Venous blood was collected for biochemistry testing.

INTERVENTIONS:
Diagnostic Test: Venous blood was collected for biochemistry testing. — For the measurement of blood tests, 10 ml of blood samples were taken from the right forearm veins with a syringe.

SUMMARY:
COVID-19 infection causes a hypersensitive immune reaction and widespread inflammation through cytokines in various organs of the body, especially the lungs.

This cytokine-mediated widespread inflammation can also affect the thyroid gland, causing thyroiditis and impaired thyroid functions.

The researchers evaluated thyroid function tests and thyroid autoantibodies in patients hospitalized for COVID-19 infection. Researchers excluded patients on intensive care therapy and patients with known thyroid disease.

The researchers examined the relationship of thyroid hormones and thyroid autoantibodies to COVID-19 disease, white blood cells, neutrophil / lymphocyte ratio, c reactive protein, fibrinogen, procalcitonin, ferritin, and D-dimer stages in these patients. Researchers compared changes in thyroid hormones and autoantibodies in people without COVID-19 infection and without thyroid disease.

DETAILED DESCRIPTION:
The coronavirus-2 (SARS-COV-2) virus, which can cause severe acute respiratory syndrome through droplet, has caused the global Coronavirus 19 (COVID-19) pandemic. COVID-19 infection can be asymptomatic as well as lead to severe illness and even death. This virus causes a hypersensitive immune reaction and varying degrees of widespread inflammation through cytokines in various organs of the body, mainly the lungs.

Cytokine-mediated widespread inflammation caused by the virus may also affect the thyroid gland and thyrocytes, causing thyroiditis and impairment of thyroid functions. Thus, it may cause changes in thyroid hormones and thyroid autoantibodies.

In study, the researchers found that in patients who were symptomatic with COVID-19 infection and who were hospitalized, thyroid function tests such as serum thyrotropin (TSH), free triiodothyronine (FT3), free thyroxine (FT4) and thyroid peroxidase antibodies (TPOAb), anti-thyroglobulin evaluated antibodies (TGAb). The investigators did not recruit patients in intensive care and patients with known thyroid disease.

Researchers looked at the association of patients' thyroid hormones and thyroid autoantibodies with white blood cells, neutrophil / lymphocyte ratio, c reactive protein, fibrinogen, procalcitonin, ferritin, D-dimer from hospital archives. The researchers determined how the thyroid hormones and autoantibodies of patients with COVID-19 infection were compared with healthy individuals without COVID-19 infection and thyroid disease.

ELIGIBILITY:
Inclusion Criteria:

* To accept research.
* Being over the age of 18.
* COVID 19 test results to be positive.
* Not taking thyroid disease medication before.
* Receiving inpatient treatment in the COVID service in the hospital.

Exclusion Criteria:

* Not accepting research.
* Be under the age of 18.
* Negative COVID 19 test results for patients.
* COVID patients treated as outpatient.
* Thyroid disease in the healthy control group.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The results of screening thyroid blood tests of healthy people without thyroid disease will be compared with the records of the COVID 19 patient group who were hospitalized and treated with no known thyroid disease.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Comparison of thyroid stimulating hormone (TSH) between groups | 90 days
  In the study, serum TSH results of the Covid patient group and non-Covid control groups were recorded and compared statistically.
Comparison of free triiodothyronine (fT3) between groups | 90 days
  In the study, serum fT3 results of the Covid patient group and non-Covid control groups were recorded and compared statistically.
Comparison of free thyroxine (fT4) between groups | 90 days
  In the study, serum fT4 results of the Covid patient group and non-Covid control groups were recorded and compared statistically.
Comparison of anti-thyroid peroxidase (Anti-TPO) between groups | 90 days
  In the study, serum anti-TPO results of the Covid patient group and non-Covid control groups were recorded and compared statistically.
Comparison of anti-thyroglobulin (Anti-Tg) between groups | 90 days
  In the study, serum anti-Tg results of the Covid patient group and non-Covid control groups were recorded and compared statistically.
White blood cells (WBC) results of Covid 19 patient group | 90 days
  In the study, serum WBC results were recorded in Covid 19 patient groups.
Neutrophil / lymphocyte ratio (N/LO) results of Covid 19 patient group | 90 days
  In the study, serum N/LO results were recorded in Covid 19 patient groups.
C-reactive protein (CRP) results of Covid 19 patient group | 90 days
  In the study, serum CRP results were recorded in Covid 19 patient groups.
Fibrinogen results of Covid 19 patient group | 90 days
  In the study, serum fibrinogen results were recorded in Covid 19 patient groups.
Procalcitonin results of Covid 19 patient group | 90 days
  In the study, serum procalcitonin results were recorded in Covid 19 patient groups.
Ferritin results of Covid 19 patient group | 90 days
  In the study, serum ferritin results were recorded in Covid 19 patient groups.
D-dimer results of Covid 19 patient group | 90 days
  In the study, serum D-dimer results were recorded in Covid 19 patient groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Sabahattin Destek, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The study will be shared when it becomes an article.

REFERENCES:
- [Background] Brancatella A, Ricci D, Viola N, Sgro D, Santini F, Latrofa F. Subacute Thyroiditis After Sars-COV-2 Infection. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa276. doi: 10.1210/clinem/dgaa276. PMID 32436948
- [Background] Caron P. Thyroid disorders and SARS-CoV-2 infection: From pathophysiological mechanism to patient management. Ann Endocrinol (Paris). 2020 Oct;81(5):507-510. doi: 10.1016/j.ando.2020.09.001. Epub 2020 Sep 18. PMID 32950466
- [Background] Mattar SAM, Koh SJQ, Rama Chandran S, Cherng BPZ. Subacute thyroiditis associated with COVID-19. BMJ Case Rep. 2020 Aug 25;13(8):e237336. doi: 10.1136/bcr-2020-237336. PMID 32843467
- [Result] van Gerwen M, Alsen M, Little C, Barlow J, Naymagon L, Tremblay D, Sinclair CF, Genden E. Outcomes of Patients With Hypothyroidism and COVID-19: A Retrospective Cohort Study. Front Endocrinol (Lausanne). 2020 Aug 18;11:565. doi: 10.3389/fendo.2020.00565. eCollection 2020. PMID 33013686